CLINICAL TRIAL: NCT04898283
Title: Prospective, Multicentre, Doubleblind, Placebo-controlled RCT to Evaluate Efficacy and Safety With SC Immunotherapy in Patients With Rhinitis/Rhinoconjunctivitis With or Without Mild to Moderate Asthma Sensitised to Grasses and Cupressaceae
Brief Title: Efficacy and Safety Evaluation of the Treatment of Allergy Against Cupressaceae and Grasses.
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Inmunotek S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DMV02-SIT-026
Record Dates: First submitted 2021-01-04; First posted 2021-05-24 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Rhinitis, Allergic; Rhinoconjunctivitis; Asthma, Allergic
Keywords: Rhinitis/ Rhinoconjunctivitis; Mild to moderate asthma; Allergy; Immunotherapy; Grass; cupressaceae
MeSH Terms: conditions — Rhinitis, Allergic; Asthma; Hypersensitivity

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, multicentre, parallel-group study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: During the trial, both the investigator and the included subjects will be unaware of the treatment each subject is receiving.
  The person in charge of data analysis will also not know the treatment assigned to each subject until the database has been closed.
  So that neither the subject nor the investigator knows what treatment each subject is receiving, all the trial medication is identical in terms of outer packaging and appearance.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 10,000 MG01 + 10,000 T521 (Experimental): 10,000 TU/mL of MG01 + 10,000 TU/mL of T521 of subcutaneous immunotherapy
  Interventions: Biological: 10,000 MG01 +10,000 T521
- 30,000 MG01 + 10,000 T521 (Experimental): 30,000 TU/mL of MG01 + 10,000 TU/mL of T521 of subcutaneous immunotherapy
  Interventions: Biological: 30,000 MG01 +10,000 T521
- Placebo subcutaneous (Placebo Comparator): The same solution and presentation as the active treatment, but without active ingredients.
  Interventions: Other: Placebo subcutaneous

INTERVENTIONS:
Biological: 10,000 MG01 +10,000 T521 — Purified and polymerized with glutaraldehyde allergen extract, from a mixture of grasses (Phleum pratense, Holcus lanatus, Poa pratensis, Festuca pratensis, Lolium perenne and Dactylis glomerata) and cupressaceae (Juniperus oxycedrus), adsorbed on aluminum hydroxide. The other ingredients are: sodium chloride (0.9%), phenol (0.4%) and water for injections
  Arms: 10,000 MG01 + 10,000 T521
Biological: 30,000 MG01 +10,000 T521 — Purified allergen extract polymerized with glutaraldehyde, from a mixture of grasses (Phleum pratense, Holcus lanatus, Poa pratensis, Festuca pratensis, Lolium perenne and Dactylis glomerata) and cupressaceae (Juniperus oxycedrus), adsorbed on aluminum hydroxide. The other ingredients are: sodium chloride (0.9%), phenol (0.4%) and water for injections.
  Arms: 30,000 MG01 + 10,000 T521
Other: Placebo subcutaneous — The same solution and presentation as the active treatment, but without active ingredients
  Arms: Placebo subcutaneous

SUMMARY:
A Randomized, Double-Blinded, Placebo-Controlled, Prospective, Multicenter Clinical Trial to Evaluate the Efficacy and Safety of Subcutaneous Immunotherapy in Patients With Rhinitis/Rhinoconjunctivitis With or Without Mild to Moderate Asthma Sensitized to cupressaceae and grasses.

DETAILED DESCRIPTION:
The multicenter study includes 180 subjects sensitised to cupressaceae and grass pollen, both male and female aged 12 to 65 years.

The double-blinded and placebo controlled treatment will last 18 months for each subject.

The primary endpoint of the trial will be the combined rhinitis/rhinoconjunctivitis symptom and medication score (RCSMS) which will be assessed using data collected in the Subject electronic Diary during the cupressaceae (January, February and March) and grass (May and June) pollen seasons.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. Aged between 12 and 65, both genders
3. Positive suggestive clinical history of intermittent or persistent moderate to severe rhinitis /rhinoconjunctivitis according to ARIA classification, with or without moderate intermittent or persistent asthma,according to GEMA 5.0, due to grass and cupressaceae pollen.
4. Subjects with a positive skin prick-test (wheal size >5 mm diameter) to a standardized mixed extract of grass pollen (Phleum pratense, Holcus lanatus, Dactylis glomerata, Poa pratensis, Festuca elatior, Lolium perenne) or to one of the molecular components of the mixture and to a cupressaceae extract. In addition, the largest diameter of the papules must be greater than or equal to that of the histamine.
5. Specific IgE > 3,5 KU/L , against grass (preferably Phleum pratense) and cupressaceae pollen (InmunoCAP® o Immulite).
6. Women of childbearing age (from menarche) must present a urine pregnancy test with a negative result at the time of joining the trial.
7. Women of childbearing potential participating in the trial, should commit to using an appropriate method of contraception. Medically acceptable methods of contraception are intrauterine devices placed at least 3 months in advance, surgical sterilization (for example, tubal ligation), barrier methods, or the use of oral contraceptives.
8. Subjects capable of complying with the dosing regimen.
9. Subjects who own a smartphone for symptom registration and medication.
10. Subjects with a negative prick test to coestational pollens. In the case specific IgE is available, the result should be <3,5 kU/L and without relevant symptomatology
11. Subjects with a negative prick test to other aeroallergens (dust mites, epitheliums and fungus). In the case specific IgE is available, the result should be <3,5 kU/L and without relevant symptomatology.

Exclusion Criteria:

1. Subjects with positive prick test to other aeroallergens except for sensitisation to epithelia with occasional exposure and symptoms.
2. Subjects with positive prick test to other aeroallergens except for sensitisation to pollen noncoseasonal with cupressus or grasses.
3. Subjects who have received prior immunotherapy in the preceding 5 years for any of the allergens tested or a cross-reactive allergen or are currently receiving immunotherapy with any allergen.
4. Subjects in which immunotherapy may be subject to an absolute general contraindication according to the criteria of the Immunotherapy Committee of the Spanish Society of Allergy and Clinical Immunology and the European Allergy and Clinical Immunology Immunotherapy Subcommittee.
5. Subjects with severe or uncontrolled intermittent or persistent asthma, with an FEV1 <70% with respect to the reference value despite adequate pharmacological treatment at the time of inclusion in the trial. Likewise, subjects with intermittent or persistent rhinitis / rhinoconjunctivitis with severe symptoms in which the suspension of oral or systemic antihistamine treatment is contraindicated.
6. Subjects who have previously had a severe secondary reaction during the prick test diagnostic skin test.
7. Subjects treated with beta-blockers.
8. Clinically unstable subjects at the time of inclusion in the trial (acute asthmatic exacerbation, respiratory infection, febrile process, acute urticaria, etc.).
9. Subjects with active chronic urticaria, severe dermographism, severe atopic dermatitis, sunburn, active psoriasis with lesions in areas where skin tests will be performed, or a history of hereditary angioedema.
10. Subjects who have any pathology in which adrenaline administration is contraindicated (hyperthyroidism, HTN, heart disease, etc.).
11. Subjects with any other disease not related to moderate rhinoconjunctivitis or asthma, but potentially serious and that may interfere with treatment and follow-up (epilepsy, psychomotor disorder, uncontrolled diabetes, malformations, multioperated patients, kidney disease,).
12. Subjects with autoimmune disease (thyroiditis, lupus, etc.), tumor diseases or with a diagnosis of immunodeficiencies.
13. Subject whose condition prevents from offering cooperation and/ or who has severe psychiatric disorders.
14. Subjects with a known allergy to components of the investigational medicinal product other than the allergen.
15. Subjects with lower respiratory diseases other than asthma such as emphysema or bronchiectasis.
16. Subjects who are direct relatives of the researchers.
17. Pregnant or lactating women.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2021-05-31 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
RCSMS: Combined Symptoms and Medication Score of rhinitis. Combined symptom and medication score in rhinitis/rhinoconjunctivitis (RCSMS) | 18 months
  Evaluation of the number of symptoms and the consumption of medication necessary for the control of such symptoms in rhinitis / rhinoconjunctivitis of each subject during the pollen season and pollen peak of cupressaceae (January, February and March) and grasses (May and June), of the groups with each other and with respect to placebo.

SECONDARY OUTCOMES:
Symptom free days | 18 months
  The number of days during the trial period that the subject was free of symptoms related to the study pathologies (both rhinitis/rhinoconjunctivitis and asthma) shall be counted for each subject.
Medication free days | 18 months
  The number of days during the trial period that the subject has not taken any medication for symptom (both rhinitis/rhinoconjunctivitis and asthma) relief shall be counted for each subject.
Symptom score in rhinitis/rhinoconjunctivitis (RSS) during pollen season and pollen peak of grasses and cupressaceae | 18 months
  The rhinitis/rhinoconjunctivitis-related symptom score shall be counted throughout the trial period for each subject.
Medication score in rhinitis/rhinoconjunctivitis (RMS) during pollen season and pollen peak of grasses and cupressaceae | 18 months
  The rhinitis/rhinoconjunctivitis-related medication score will be counted throughout the trial period for each subject.
Combined symptom and medication score (ACSMS) during pollen season and pollen peak of grasses and cupressaceae | 18 months
  The combined asthma-related symptom score (ASS) and asthma-related medication score (AMS) shall be counted throughout the trial period for each subject.
  The ACSMS shall range from 0 to 6.
Asthma symptom score (ASS) during pollen season and pollen peak of grasses and cupressaceae | 18 months
  The asthma-related symptom score shall be counted throughout the trial period for each subject. The symptoms are as follows: coughing, wheezing or whistling, choking or suffocating sensation, chest tightness
  The assessment criteria for each symptom shall be as follows:
  0 = No symptoms (no obvious symptoms).
  1. = Mild (trivial; the symptom is clearly present but not bothersome).
  2. = Moderate (annoying, but not disabling or intolerable).
  3. = Severe (disabling and/or intolerable). The asthma symptom score (ASS) will be the sum of the 4 asthma symptoms divided by 4. The final score will vary from 0 to 3.
Asthma Medication Score (AMS) during pollen season and pollen peak of grasses and cupressaceae | 18 months
  The asthma-related medication score will be counted throughout the trial period for each subject. The medication will be scored based on the therapeutic step in which the drugs are included in the GEMA 5.0 and GINA 2020 guidelines. The scoring approach is detailed in the article entitled 'Combination of Allergic Asthma Symptom and Medication Scores in Allergen Immunotherapy Trials: A Proposal'
Asthma and rhinitis/rhinoconjunctivitis symptom score (ARSS) during pollen season and pollen peak of grasses and cupressaceae | 18 months
  The asthma-related (ASS) and rhinitis/rhinoconjunctivitis (RSS) symptom scores shall be counted throughout the trial period for each subject.
  The ARSS shall range from 0 to 6.
Asthma and rhinitis/rhinoconjunctivitis medication score (ARMS) during pollen season and pollen peak of grasses and cupressaceae | 18 months
  The asthma-related medication score (AMS) and rhinitis/rhinoconjunctivitis score (RMS) shall be counted throughout the trial period for each subject.
  The ARMS shall range from 0 to 6.
Combined symptom and medication score in asthma and rhinitis/rhinoconjunctivitis (ARCSMS) during pollen season and pollen peak of grasses and cupressaceae | 18 months
  The combined asthma-related symptom and medication score (ACSMS) and rhinitis/rhinoconjunctivitis (RCSMS) shall be counted throughout the trial period for each subject.
  The ARCSMS shall range from 0 to 12.
Asthmatic exacerbations | 18 months
  Time to first occurrence of asthmatic exacerbation, number, duration and severity will be analysed.
Visual Analogue Scale (VAS) | 18 months
  Visual Analogue Scale in which the subject has to indicate in a straight line of 10cm how he/she feels regarding to his allergy symptoms. Being left side (0) = very bad and right side (10) = very well
Immunological parameters | 18 months
  Total IgE, specific IgE and specific IgG4 are analysed during screening and final visit.
  The determination of grasses shall be carried out on Phleum pratense. The determination of immunological parameters shall be carried out by analysis of the whole or total extract and not by molecular components.
Quality of life associated with asthma (ACQ-6) | 18 months
  The quality of life associated with asthma will be measured following the ACQ questionnaire.
  The ACQ questionnaire consists of 6 questions (ACQ-6). In questions 1-6, patients recall their experience during the last 7 days and answer using a scale of 7 points (from 0 = fully controlled to 6 = extremely poorly controlled). The questionnaire score is the mean of the 6 responses (ACQ-6).
  The interpretation of the scores is as follows:
  Less than or equal to 0.75: Adequate control of asthma From 0.75 to 1.50: Partially controlled asthma More than 1.50: Inadequate asthma control
Quality of life associated with rhinitis (ESPRINT-15) | 18 months
  The quality of life associated with rhinitis will be measured following the test ESPRINT-15.
  The scoring of the questionnaire will be carried out as follows: The global sum of the scores (ranging from "0 = nothing has bothered me" to "6 = it has bothered me a lot") of the 14 items plus the score given in the general questionnaire (ranging from "0 = Excellent" to "4 = Bad"). This sum is divided by the total number of items (15 items).
  The interpretation of the scores is between 0 (low impact) and 6 (high impact).
Health resource consumption | 18 months
  Counting the Health resource consumption related to the study pathology: visits to specialists, telephone calls, test and analyses.
  Recording of health resource consumption will be carried out at all study visits, from screening to final visit or additional final visit, if applicable.
Safety parameters | 18 months
  Number of participants with treatment-related adverse events as assessed by T521+MG01-SIT026.
  Comparison between the beginning and end of the trial and among active groups and placebo

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Ojeda, MD, Study Director — Clínica privada Dres Ojeda
Locations (27):
- Spain (27):
  - Hospital Recoletas Felipe Ii, Valladolid, Castille and León
  - Cedt de Tarancón, Tarancón, Cuenca
  - Hospital Universitario Principe de Asturias, Alcalá de Henares, Madrid
  - Hospital U. Fundación Alcorcón, Alcorcón, Madrid
  - Hospital Cruz Roja Madrid, Madrid, Madrid
  - Clínica Privada Dres Ojeda, Madrid, Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Clínica Privada Murcia, Murcia, Murcia
  - Hospital Nuestra Señora de Sonsoles, Ávila
  - Fundación Hospital Sant Pere Claver, Barcelona
  - Clínica privada Burgos, Burgos
  - Hospital Universitario de Burgos, Burgos
  - Hospital General de Villalba, Collado Villalba
  - Clinica privada, León
  - Clínica Subiza, Madrid
  - Hospital Carlos III (antiguo CAP José Marva), Madrid
  - Clínica Privada, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Infanta Elena, Madrid
  - Centro médico Saluddia, Madrid
  - Centro Médico Iza (Clínica Privada Madrid), Madrid
  - Consulta Privada, Palencia
  - Hospital Clínico de Salamanca, Salamanca
  - Hospital General Universitario de Segovia, Segovia
  - Clinica Privada Soria, Soria
  - Clínica Privada, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guzman-Fulgencio M, Caballero R, Lara B, Mena M, Tejera M, Sastre A, Subiza JL, Fernandez-Caldas E, Casanovas M. Safety of immunotherapy with glutaraldehyde modified allergen extracts in children and adults. Allergol Immunopathol (Madr). 2017 Mar-Apr;45(2):198-207. doi: 10.1016/j.aller.2016.08.008. Epub 2016 Dec 7. PMID 27939406
- [Background] Caballero R, Grau A, Javaloyes G, Del Pozo S, Leon MA, Romero M, Casanovas M. Combination of Allergic Asthma Symptom and Medication Scores in Allergen Immunotherapy Trials: A Proposal. Int Arch Allergy Immunol. 2021;182(7):571-573. doi: 10.1159/000513543. Epub 2021 Jan 26. No abstract available. PMID 33498057